CLINICAL TRIAL: NCT00365222
Title: Phase II Study of Dose Intensive Temozolomide in Elderly Adults With Newly Diagnosed Glioblastoma
Brief Title: Phase II Study of Temozolomide in Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Study Closure
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Marc Chamberlain, M.D., H. Lee Moffitt Cancer Center and Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14714
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Temozolomide; Temodar; Glioblastoma; Gliosarcoma; Brain Tumor; Quality of Life; Neurological
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Neurologic Manifestations | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — temozolomide 75 mg/m2 /d
  Other Names: Temodar

SUMMARY:
A single arm Phase 2 trial with the study drug temozolomide (temodar) for newly diagnosed glioblastoma in elderly patients (defined as greater than or equal to 70 years old). Following surgical resection, and confirmation of glioblastoma, patients will proceed to primary chemotherapy with temozolomide (temodar). Temodar is given for 42 consecutive days on and 14 days off occurring every 56 days.

Procedures prior to initial study treatment (<14 Days) are: Neurological/Oncological History, Neurological Examination, Height, Weight, and Body Surface Area, Performance Status, Quality Of Life FACT-BR, Labs, MGMT tissue analysis, and Cranial CT/MRI with and without contrast.

The same procedures are repeated on Day 1 of each treatment cycle with the addition of an adverse event assessment. And the off study procedures for patients are performance status, Quality Of Life FACT-BR, MGMT tissue analysis, and cranial CT/MRI with and without contrast.

Patients may continue with each temodar daily dose therapy if clinical and neuroradiographical exams are stable or improving.

DETAILED DESCRIPTION:
A single arm Phase 2 trial with the study drug temozolomide (temodar) for newly diagnosed glioblastoma in elderly patients (defined as greater than or equal to 70 years old). Temozolomide will be administered orally (a capsule) at approximately the same time daily (bedtime) for 42 days on and then 14 days off; cycles may be repeated every 56 days. Complete blood counts will be obtained bi-weekly, evaluations monthly and MRI's every 2 months after a cycle of therapy.

Procedures prior to initial study treatment (<14 Days) are: Neurological/Oncological History, Neurological Examination, Height, Weight, and Body Surface Area, Performance Status, Quality Of Life FACT-BR, Labs, MGMT tissue analysis, and Cranial CT/MRI with and without contrast (all disease found at staging must be followed using the same modality used at Pre-treatment. Tumor assessments are to be repeated every 56 days thereafter until progression). The same procedures are repeated on Day 1 of each treatment cycle with the addition of an adverse event assessment.

Patients may continue on therapy unless one of the following occurs:

* Documented or clinical progressive disease at any time
* Unacceptable toxicity
* Treatment delay of > 2 weeks for any reason
* Study data or other data indicate that the study treatment is not beneficial for the patients; defined as at least one response in the first 12 patients within each tumor histology strata
* Non-compliance by the patient with protocol requirements (follow-up, treatment, administration of disallowed therapy)
* Changes in medical status of the patient such that the patient no longer meets eligibility requirements (leptomeningeal spread, change in mental competency) or the investigator believes that patient safety will be compromised.
* Patient withdrawal of consent for treatment
* Occurrence of one toxic death

Patients with CR, PR, or stable disease (SD) will be treated for a minimum of 3 cycles [6 months] or until disease progression. For patients responding to treatment, continuation of therapy beyond 3 cycles is at the discretion of the investigator. Response parameters will include the MacDonald criteria for evaluating brain tumors. Response is measured by a reduction in tumor size.

After cessation of protocol therapy, patients will continue to be followed for survival at 2-month intervals for up to three years from start of treatment. And the off study procedures for patients are performance status, Quality Of Life FACT-BR, MGMT tissue analysis, and cranial CT/MRI with and without contrast.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological documented glioblastoma or gliosarcoma. All patients must have had prior pathologic confirmation of tumor histology.
* Patients must be > than or equal to 70 years old.
* Patients must have a Karnofsky performance status of > 50.
* Nonmeasurable disease or measurable disease per MacDonald criteria
* Patients must have a predicted life expectancy of at least 12 weeks.
* Required initial laboratory data: ANC >1,500, Platelets >100,000, Serum Creatinine <2.0, Serum Bilirubin <2.0, and AST/ALT <3x normal
* Patients must sign and date an IRB approved informed consent form stating he or she is aware of the neoplastic nature of the disease. Patient must willingly provide written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts. (Human protection committee approval of this protocol and consent form is required).
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests and accessible for follow-up.
* Patients must have been previously treated with surgery.
* No prior adjuvant or salvage chemotherapy regimen is permitted.
* Prior radiotherapy is not permitted.

Exclusion Criteria:

* Patients have evidence of leptomeningeal spread of disease.
* Patients having been treated with prior chemotherapy or radiotherapy.
* Patients with a second active malignancy or diagnosis of other cancer within -3 years of enrollment, except for surgically cured basal cell carcinoma, or in situ carcinoma of the cervix.
* Mentally incapacitated patients or psychiatric illness that would prevent the patient from giving informed consent.
* Patients with poorly controlled diabetes, hepatitis infection, uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, and myocardial infarction within the previous six months, or serious uncontrolled cardiac arrhythmia.
* Known to be HIV positive or to have an AIDS-related illness.
* Patients with an active infection that is not adequately controlled with antibiotics.
* Patients with other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Patients with a known sensitivity to any of the products to be administered during treatment.
* Patients currently enrolled in another clinical trial or patients who have participated in a trial of an investigational device or drug within the last 30 days.
* Patients previously treated with temozolomide.
* Concurrent radiotherapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluate overall survival | dependent upon results

SECONDARY OUTCOMES:
Progression-free survival at six and nine months | 9 months
Response rate measured by a reduction in tumor size | 9 months
Frequency and severity of adverse events | 9 months
Quality of life measured at each cycle utilizing the QOL FACT-BR | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Chamberlain, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org